CLINICAL TRIAL: NCT01797549
Title: Detection of Hemodynamic Changes in TBI Population With Functional Near Infrared Spectroscopy
Status: Completed | Type: Observational
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: Center for Neuroscience and Regenerative Medicine (CNRM) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ramon Diaz-Arrastia, Director of Clinical Research, Uniformed Services University of the Health Sciences
Other Study IDs: 0189AP
Record Dates: First submitted 2013-02-07; First posted 2013-02-22 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury; functional near infrared spectroscopy
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- History of having sustained TBI: Males and females between 18 and 60 years who have a diagnosis of TBI
- Control group: Control group with no history of TBI or concussion. Gender and age matched non-TBI volunteers

SUMMARY:
The goal of this project is to develop a test to assess frontal lobe function using a rapid, inexpensive, objective, and standardized method, without the need for expertise in cognitive test administration. Such methods would be particularly helpful in traumatic brain injury (TBI), where objective measures are needed, and would greatly expand the capacity to make such assessments in clinical practice and research.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, write, speak and understand English
* history of having sustained a TBI prior to enrollment. Evidence will be any one of the following 3 criteria:

  1. GCS 3 - 12
  2. Post-traumatic amnesia > 24 hours
  3. TBI-related abnormality on neuroimaging (either CT or MRI). (Some missing information about the initial injury (i.e. documentation of initial GCS) is not necessarily exclusionary if the bulk of the available history is indicative that the patient suffered a TBI and meets the inclusion criteria)

Exclusion Criteria:

* Multiple sclerosis, pre- or co-existing
* Stroke (other than stroke at the time of TBI)
* Pre-existing developmental disorder
* Pre-existing epilepsy
* Pre-existing major depressive disorder
* Pre-existing schizophrenia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Males and females (military health care beneficiaries and non military health care beneficiaries) age between 18 and 60 years who have a diagnosis of moderate or severe traumatic brain injury as well as age, gender, education matched non-TBI volunteers.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Measure of hemodynamic response function | Two years
  In two population groups: TBI and non TBI, we will determine normative data for the cognitive parametric experiment by measuring the local hemodynamic response function with functional near infrared spectroscopy

SECONDARY OUTCOMES:
Measure of the degree of impairment | Two years
  Determine the relationship between hemodynamic response as measured by fNIRS and measures of neuropsychological and behavioral functioning obtained using measures from the NINDS Common Data Elements.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Neuroscience and Regenerative Medicine (CNRM), Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chernomordik V, Amyot F, Kenney K, Wassermann E, Diaz-Arrastia R, Gandjbakhche A. Abnormality of low frequency cerebral hemodynamics oscillations in TBI population. Brain Res. 2016 May 15;1639:194-9. doi: 10.1016/j.brainres.2016.02.018. Epub 2016 Mar 17. PMID 26996413